CLINICAL TRIAL: NCT03114475
Title: Evaluation of Enamel Resistance to White Spot Lesion Formation Around Orthodontic Brackets After CO2 Laser Irradiation: A Randomized Controlled Clinical Trial
Brief Title: Effect of CO2 Laser on Enamel White Spot Lesion Formation Around Orthodontic Brackets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: UDDS-Ortho-01-2017
Record Dates: First submitted 2017-04-11; First posted 2017-04-14 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: White Spot Lesion

STUDY DESIGN:
Intervention Model Description: Split mouth design, the mouth will be split into four quadrants. Two quadrants will receive the active treatment, whereas the opposing two quadrants will receive the placebo.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The non-irradiated side of the mouth will receive a placebo light (i.e. not the laser beam).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CO2 Laser Irradiation (Experimental): This group of patients will be treated by splitting the dental arches into four quadrants: upper right, upper left, lower right and lower left. Two quadrants will receive the CO2 laser irradiation whereas the remaining two quadrants will receive no treatment (i.e. the placebo light).
  Interventions: Radiation: CO2 laser irradiation
- Placebo (Placebo Comparator): A placebo light will be used as if the patient is irradiated with the laser beam.
  Interventions: Other: Placebo

INTERVENTIONS:
Radiation: CO2 laser irradiation — CO2 laser irradiation will be applied onto the enamel surrounding the orthodontic bracket
  Arms: CO2 Laser Irradiation
Other: Placebo — No irradiation is going to be applied in the intervention. Just a red light will be used as placebo.
  Arms: Placebo

SUMMARY:
This study aims to evaluate the clinical effect of CO2 laser on enamel resistance to white spot lesions formation around orthodontic brackets.

25 patients needing fixed orthodontic treatment will participate in the study, the CO2 laser will be applied in a split mouth design around orthodontic brackets in two contrast quarters of mouth in every patient and the other quarters will serve as a control. The white spot lesion formation will be monitored around the brackets during the orthodontic treatment after four and twelve weeks of irradiation with laser.

DETAILED DESCRIPTION:
Prior to enrollment of each subject into the study, they will be examined completely to determine the orthodontic treatment plan. The operator will inform them about the aim of the study and ask them to provide a written informed consent.

Before brackets' bonding (T0) the operator will evaluate with intraoral clinical examination and take intraoral photographs and evaluate with DIAGNOdent. Then after brackets' placement on teeth, the CO2 laser will be applied to the area of enamel about 2 mm of width around orthodontic brackets in a split mouth design. To blind the intervention sides on patients the control sides will receive nontherapeutic light.

Then intraoral photographs will be taken and the teeth will be assessed with DIAGNOdent (T1).

All patients will be trained to brush their teeth with a tooth paste containing 1100 ppm of fluoride twice a day. After 4 weeks of irradiation (T2) the patients will be examined for white spot lesions formation by clinical examination using Geiger index, photographic examination using AutoCAD 2009 evaluating formation and area percentage of white spot lesions, and the degree of demineralization will be assessed with DIAGNOdent. The all exams will also be done after 12 weeks of irradiation (T3).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with permanent occlusion at age 15-25 years.
* No previous orthodontic treatment
* Good oral hygiene
* Need to orthodontic treatment with fixed appliances

Exclusion Criteria:

* Patients with systemic diseases or syndromes
* Patients with existence of enamel fluorosis
* Patients with existence of amelogenesis imperfecta or hypocalcified enamel
* Patients with existence of restorations or crowns or carious lesions on the labial surfaces of teeth.
* Patients who received fluoride treatment within the last three months prior to being enrolled in the study.

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in White Formation Status we will evaluate the degree of demineralization by DIAGNOdent Pen around the orthodontic brackets. | The status of white spot formation will be judged at 10 minutes before taking the impressions (T0), five minutes following brackets' placement and irradiation (T1), at four weeks after laser irradiation (T2) and at twelve weeks after irradiation (T3)
  This will depend on the presence or absence of white spot formation assessed clinically.
Change in the Extent of White Spot Formation | Extent of white spot formation will be measured 10 minutes before taking the impressions (T0), five minutes following brackets' placement and irradiation (T1), at four weeks after laser irradiation (T2) and at twelve weeks after laser irradiation (T3)
  This will be assessed clinically using Geiger index (Step 1: no white spot lesions, Step 2: the white spot lesion is less than the third of the tooth surface area, Step 3: the white spot lesion is more than the third of the tooth surface area, Step 4: severe white spot lesions and caries)
Change in the Percentage of White Spot Lesion Area | Percentage of white spot lesion area will be assessed at 10 minutes before taking the impressions (T0), five minutes following brackets' placement and irradiation (T1), at four weeks after irradiation (T2) and at twelve weeks after irradiation (T3)
  This will be assessed using digital images.The percentage of white spot lesion area to the area of the labial surface of the tooth on digital images will be calculated using AutoCAD 2013 program.
Change in the degree of demineralization | The degree of demineralization will be evaluated at: t 10 minutes before taking the impressions (T0), five minutes following brackets' placement and irradiation (T1), at four weeks after irradiation (T2) and at twelve weeks after irradiation (T3)
  The degree of demineralization will be evaluated by DIAGNOdent Pen around the orthodontic brackets.

CONTACTS AND LOCATIONS:
Overall Officials: Tuqa Raghis, DDS, Principal Investigator — MSc student, Department of Orthodontics, University of Damascus Dental School; Ghiath Mahmoud, DDS MSc PhD, Study Director — Senior Lecturer in Orthodontics, Department of Orthodontics, University of Damascus Dental School, Damascus, Syria
Locations (2):
- Syria (2):
  - Department of Orthodontics, University of Damascus Dental School, Damascus
  - Higher Institution for Laser Research and Applications, Damascus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Esteves-Oliveira M, Zezell DM, Meister J, Franzen R, Stanzel S, Lampert F, Eduardo CP, Apel C. CO2 Laser (10.6 microm) parameters for caries prevention in dental enamel. Caries Res. 2009;43(4):261-8. doi: 10.1159/000217858. Epub 2009 May 8. PMID 19439947
- [Background] Esteves-Oliveira M, Pasaporti C, Heussen N, Eduardo CP, Lampert F, Apel C. Prevention of toothbrushing abrasion of acid-softened enamel by CO(2) laser irradiation. J Dent. 2011 Sep;39(9):604-11. doi: 10.1016/j.jdent.2011.06.007. Epub 2011 Jun 30. PMID 21741428
- [Background] Gomez J. Detection and diagnosis of the early caries lesion. BMC Oral Health. 2015;15 Suppl 1(Suppl 1):S3. doi: 10.1186/1472-6831-15-S1-S3. Epub 2015 Sep 15. PMID 26392124
- [Background] Miresmaeili A, Farhadian N, Rezaei-soufi L, Saharkhizan M, Veisi M. Effect of carbon dioxide laser irradiation on enamel surface microhardness around orthodontic brackets. Am J Orthod Dentofacial Orthop. 2014 Aug;146(2):161-5. doi: 10.1016/j.ajodo.2014.04.023. PMID 25085298
- [Background] Rechmann P, Fried D, Le CQ, Nelson G, Rapozo-Hilo M, Rechmann BM, Featherstone JD. Caries inhibition in vital teeth using 9.6-mum CO2-laser irradiation. J Biomed Opt. 2011 Jul;16(7):071405. doi: 10.1117/1.3564908. PMID 21806251
- [Background] Rechmann P, Charland DA, Rechmann BM, Le CQ, Featherstone JD. In-vivo occlusal caries prevention by pulsed CO2 -laser and fluoride varnish treatment--a clinical pilot study. Lasers Surg Med. 2013 Jul;45(5):302-10. doi: 10.1002/lsm.22141. Epub 2013 Jun 4. PMID 23737079
- [Background] Seino PY, Freitas PM, Marques MM, de Souza Almeida FC, Botta SB, Moreira MS. Influence of CO2 (10.6 mum) and Nd:YAG laser irradiation on the prevention of enamel caries around orthodontic brackets. Lasers Med Sci. 2015 Feb;30(2):611-6. doi: 10.1007/s10103-013-1380-8. Epub 2013 Jun 30. PMID 23812850
- [Background] Souza-Gabriel AE, Colucci V, Turssi CP, Serra MC, Corona SA. Microhardness and SEM after CO(2) laser irradiation or fluoride treatment in human and bovine enamel. Microsc Res Tech. 2010 Oct;73(11):1030-5. doi: 10.1002/jemt.20827. PMID 20146349
- [Background] Stangler LP, Romano FL, Shirozaki MU, Galo R, Afonso AM, Borsatto MC, Matsumoto MA. Microhardness of enamel adjacent to orthodontic brackets after CO2 laser irradiation and fluoride application. Braz Dent J. 2013 Sep-Oct;24(5):508-12. doi: 10.1590/0103-6440201302292. PMID 24474294
- [Background] Steiner-Oliveira C, Rodrigues LK, Soares LE, Martin AA, Zezell DM, Nobre-dos-Santos M. Chemical, morphological and thermal effects of 10.6-microm CO2 laser on the inhibition of enamel demineralization. Dent Mater J. 2006 Sep;25(3):455-62. doi: 10.4012/dmj.25.455. PMID 17076314
- [Derived] Raghis T, Mahmoud G, Abdullah A, Hamadah O. Enamel resistance to demineralisation around orthodontic brackets after CO2 laser irradiation: a randomised clinical trial. J Orthod. 2018 Dec;45(4):234-242. doi: 10.1080/14653125.2018.1504410. Epub 2018 Aug 2. PMID 30071781